CLINICAL TRIAL: NCT02889510
Title: Multicentre Randomized Double Blind, Crossover, Placebo Controlled Clinical Trial to Evaluate the Effect of Liraglutide on Lung Function in Patients With Type 2 Diabetes Mellitus (LIRALUNG Study)
Brief Title: Study to Assess the Efficacy of Liraglutide in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lecube, Albert, M.D. (Individual)
Collaborators: Dynamic Solutions (Industry); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LIRALUNG
Record Dates: First submitted 2016-08-25; First posted 2016-09-05 (Estimated); Results first posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; liraglutide; lung function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide (Other): 7-week subcutaneous liraglutide treatment once daily
  Interventions: Drug: liraglutide
- placebo (Other): 7-week subcutaneous placebo treatment once daily.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 7-week subcutaneous liraglutide once daily
  Arms: liraglutide
Drug: placebo — 7-week subcutaneous placebo once daily
  Arms: placebo

SUMMARY:
Type 2 diabetes (T2DM) is related to reduced pulmonary function. As experimental studies with glucagon-like peptide 1 (GLP-1) have shown an increase in pulmonary surfactant secretion, and the GLP-1 receptor has been found in significant amounts in the lung, it could be hypothesized that the treatment with liraglutide (a GL-1 agonist) will improve this reduced pulmonary function

DETAILED DESCRIPTION:
There is growing evidence to suggest an association between type 2 diabetes and impaired pulmonary function. In this regard, several cross-sectional studies have appeared showing decreased indices of forced expiration, lung volume and diffusion capacity as the main lung dysfunctions detected in type 2 diabetic populations. In fact, diabetes is frequently co-morbid with chronic obstructive pulmonary disease, and data from the Atherosclerosis Risk in Communities Study showed a faster pulmonary function decline in type 2 diabetic patients than in other participants. This is important because the reduction of FEV1 has been demonstrated an independent cause of mortality in diabetic patients.

Interestingly, lung function measures start to decrease several years before the diagnosis of diabetes. In this regard an investigation found that insulin resistance is an independent determinant of pulmonary function in non-diabetic morbidly obese women. In addition, the results suggest that the metabolic pathways related to insulin resistance are crucial in initiating lung abnormalities in type 2 diabetic patients.

The reasons for the association between respiratory disease and diabetes are unclear. However, the relationship between type 2 diabetes and muscle strength, the impairment in lung elastic properties, and the presence of a low-grade chronic inflammation state are involved. In supporting these findings, thickening of the alveolar epithelia and pulmonary capillary basal lamina, fibrosis, centrilobular emphysema, and pulmonary microangiopathy have been detected in autopsies of diabetic patients. In addition, defects in the bronchiolar surfactant layer, which is involved in maintaining airway stability and diameter, may also be considered a contributing factor to the impairment of airway calibre regulation in diabetic patients. When the alveolocapillary barrier is damaged, surfactant proteins leak into the bloodstream. A recent population-based random sample study has described how increased circulating levels of surfactant protein A, the major surfactant-associated protein, were associated with altered glucose tolerance and insulin resistance. Therefore, surfactant defects in diabetic individuals may also lead to an increase in airway resistance and to a reduction in ventilatory patterns as observed in our studies. In addition, as experimental studies have shown that glucagon-like peptide 1 plays a role in the stimulation of surfactant production, its underlying deficit in type 2 diabetes could also enhance the airway resistance observed in these patients. However, the beneficial effects on pulmonary function using incretin-based therapies remain to be elucidated.

Clinical trial study hypothesis is that treatment with an incretin mimetic such as liraglutide may ameliorate lung function parameters in type 2 diabetics patients, independently of weight reduction. This hypothesis is based on the following factors:

1. - There is growing evidence to suggest an association between type 2 diabetes and impaired pulmonary function.
2. - In patients with type 2 diabetes, the incretin effect is severely reduced or absent, contributing to the reduced lung function parameters observed in type 2 diabetic patients.
3. - GLP-1 stimulates surfactant production in "in vitro" studies and, in consequence, the increase in surfactant production induced by liraglutide could be the main factor involved in the respiratory improvement.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Subjects between 40 and 65 years old. Diagnosis of type 2 diabetes mellitus with more than 5 years of evolution of disease.
* Metformin (alone or in combination with sulfonylurea and / or insulin and / or thiazolidinediones) at a stable dose for at least the past 3 months.
* HbA1c ≥ 7,0 y ≤ 9,0 %.
* BMI between 30 and 40 kg / m2.
* No pulmonary disease (COPD, asthma, fibrosis, etc) known.
* Baseline FEV1 decline of equal or greater than 10% in the percentage of the theoretical value.
* Chest radiography without significant changes in the lung parenchyma

Exclusion Criteria:

* Type 1 diabetes mellitus
* Treatment with inhibitors of dipeptidyl peptidase 4 glitazones and / or
* SGLT2 inhibitors.
* Active and former smokers for less than five years ago smoking.
* Chronic obstructive pulmonary disease.
* Respiratory sleep disorders that require treatment with continuous positive pressure in the airway.
* Asthma treatment with bronchodilators.
* Previous bariatric surgery.
* Cardiovascular disease, heart failure and / or stroke.
* Pathology of the chest wall.
* Serum creatinine> 1.7 mg / dl.
* Abnormal results in liver function test (Alanine transaminase/ Aspartate Aminotransferase greater than twice the upper limit of normal).
* History of acute or chronic pancreatitis.
* Personal or family history of medullary thyroid cancer or Multiple
* Endocrine Neoplasia (MEN ) type 2.
* Active neoplasms or neoplastic patients considered disease-free history from less than 5 years ago.
* Women of childbearing age who are pregnant (positive pregnancy test within 14 days before the start of treatment) or intend to get pregnant.
* Lactating women.
* Women of childbearing potential not using adequate contraception (such as oral contraceptives, intrauterine device or barrier method of birth control along with spermicide or surgical sterilization) or unwilling to use during the study (as required by local laws or practices).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lecube, PhD, Study Director — Hospital Universitari Arnau de Vilanova de Lleida
Locations (6):
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d´Hebrón, Barcelona
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis TM, Knuiman M, Kendall P, Vu H, Davis WA. Reduced pulmonary function and its associations in type 2 diabetes: the Fremantle Diabetes Study. Diabetes Res Clin Pract. 2000 Oct;50(2):153-9. doi: 10.1016/s0168-8227(00)00166-2. PMID 10960726
- [Background] Yeh HC, Punjabi NM, Wang NY, Pankow JS, Duncan BB, Cox CE, Selvin E, Brancati FL. Cross-sectional and prospective study of lung function in adults with type 2 diabetes: the Atherosclerosis Risk in Communities (ARIC) study. Diabetes Care. 2008 Apr;31(4):741-6. doi: 10.2337/dc07-1464. Epub 2007 Dec 4. PMID 18056886
- [Background] Vara E, Arias-Diaz J, Garcia C, Balibrea JL, Blazquez E. Glucagon-like peptide-1(7-36) amide stimulates surfactant secretion in human type II pneumocytes. Am J Respir Crit Care Med. 2001 Mar;163(4):840-6. doi: 10.1164/ajrccm.163.4.9912132. PMID 11282754
- [Background] Lecube A, Sampol G, Munoz X, Lloberes P, Hernandez C, Simo R. Insulin resistance is related to impaired lung function in morbidly obese women: a case-control study. Diabetes Metab Res Rev. 2010 Nov;26(8):639-45. doi: 10.1002/dmrr.1131. Epub 2010 Sep 29. PMID 20882512
- [Background] Lecube A, Sampol G, Munoz X, Hernandez C, Mesa J, Simo R. Type 2 diabetes impairs pulmonary function in morbidly obese women: a case-control study. Diabetologia. 2010 Jun;53(6):1210-6. doi: 10.1007/s00125-010-1700-5. Epub 2010 Mar 9. PMID 20217039
- [Background] Lecube A, Sampol G, Lloberes P, Romero O, Mesa J, Hernandez C, Simo R. Diabetes is an independent risk factor for severe nocturnal hypoxemia in obese patients. A case-control study. PLoS One. 2009;4(3):e4692. doi: 10.1371/journal.pone.0004692. Epub 2009 Mar 5. PMID 19262746
- [Background] Fernandez-Real JM, Chico B, Shiratori M, Nara Y, Takahashi H, Ricart W. Circulating surfactant protein A (SP-A), a marker of lung injury, is associated with insulin resistance. Diabetes Care. 2008 May;31(5):958-63. doi: 10.2337/dc07-2173. Epub 2008 Feb 19. PMID 18285549
- [Background] Mannino DM, Thorn D, Swensen A, Holguin F. Prevalence and outcomes of diabetes, hypertension and cardiovascular disease in COPD. Eur Respir J. 2008 Oct;32(4):962-9. doi: 10.1183/09031936.00012408. Epub 2008 Jun 25. PMID 18579551
- [Background] Davis WA, Knuiman M, Kendall P, Grange V, Davis TM; Fremantle Diabetes Study. Glycemic exposure is associated with reduced pulmonary function in type 2 diabetes: the Fremantle Diabetes Study. Diabetes Care. 2004 Mar;27(3):752-7. doi: 10.2337/diacare.27.3.752. PMID 14988297
- [Background] Nicolaie T, Zavoianu C, Nuta P. Pulmonary involvement in diabetes mellitus. Rom J Intern Med. 2003;41(4):365-74. PMID 15526520
- [Derived] Lopez-Cano C, Ciudin A, Sanchez E, Tinahones FJ, Barbe F, Dalmases M, Garcia-Ramirez M, Soto A, Gaeta AM, Pellitero S, Marti R, Hernandez C, Simo R, Lecube A. Liraglutide Improves Forced Vital Capacity in Individuals With Type 2 Diabetes: Data From the Randomized Crossover LIRALUNG Study. Diabetes. 2022 Feb 1;71(2):315-320. doi: 10.2337/db21-0688. PMID 34737187

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: It is a cross-over study so patients are in both arms if they complete all the study. The order of the treatment received depends on the group assigned:
  A= treatment with subcutaneus liraglutide for 7 weeks once daily followed by treatment with subcutaneus placebo for 7 weeks B= treatment with subcutaneus placebo for 7 weeks once daily followed by treatment with subcutaneus liraglutide for 7 weeks
  76 participants were enrolled in the study but only 72 started the treatment.
Groups:
- Liraglutide First, Then Placebo: treatment with subcutaneus liraglutide for 7 weeks once daily followed by treatment with subcutaneus placebo for 7 weeks
- Placebo First, Then Liraglutide: treatment with subcutaneus placebo for 7 weeks once daily followed by treatment with subcutaneus liraglutide for 7 weeks
Period: Overall Study
Arm/Group | Liraglutide First, Then Placebo | Placebo First, Then Liraglutide
Started | 35 | 37
Completed | 27 | 32
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 73
  Arab | 1
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 76
Never smokers [Count of Participants; unit: Participants] | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Two arms.
  kg/m^2
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 34.7 (4.2)
    Placebo first,then liraglutide: number analyzed (Participants) | 38
    Placebo first,then liraglutide | 35 (4.4)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Two arms.
  mmHg
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 146.9 (17.3)
    Placebo first,then liraglutide: number analyzed (Participants) | 38
    Placebo first,then liraglutide | 145.2 (19.8)
Fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] — Population: Two arms.
  mmol/L
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 11.0 (3.5)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 10.9 (4.0)
Glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 8.3 (1.1)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 7.9 (0.9)
Glycated hemoglobin (HbA1c) [Median (Standard Deviation); unit: mmol/mol] — Population: Two arms.
  mmol/mol
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 67.2 (12.1)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 63.7 (10.5)
Forced expiratory volume in 1s (FEV1) [Mean (Standard Deviation); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 81.1 (12.1)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 77.8 (12.1)
Forced vital capacity (FVC) [Mean (Standard Deviation); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 81.9 (18.8)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 79.6 (12.6)
Maximum mid-expiratory flow (FEF25-75) [Mean (Standard Deviation); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 79.2 (27.2)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 70.1 (28.9)
Peak expiratory flow (PEF) [Mean (Standard Deviation); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 80.7 (27.2)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 80.7 (27.8)
FEV1/FVC [Mean (Inter-Quartile Range); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 81.6 [77.1 to 89]
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 82.3 [77.6 to 90]
Non obstructive ventilatory defect (VD) [Mean (Standard Deviation); unit: %] — Population: Two arms.
  %
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 27 (37.5)
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 25 (38.4)
Surfactant A protein [Median (Inter-Quartile Range); unit: ng/ml] — Population: Two arms.
  ng/ml
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 35.6 [19.4 to 46.9]
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 34.2 [20.5 to 46.8]
Surfactant D protein [Median (Inter-Quartile Range); unit: ng/ml] — Population: Two arms
  ng/ml
    Liraglutide first, then placebo: number analyzed (Participants) | 38
    Liraglutide first, then placebo | 196.5 [128.3 to 271.5]
    Placebo first, then liraglutide: number analyzed (Participants) | 38
    Placebo first, then liraglutide | 184.2 [118.3 to 287.3]

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Forced Expiratory Volume in 1 Second (FEV1)
Description: Changes from baseline on measurements of respiratory function defined by forced expiratory volume in 1 second (FEV1).
  Mean difference between 7 weeks after treatment visit and baseline visit is registered.
Time Frame: 7 weeks
Population: 59 patients ended the period of 7 weeks of liraglutide treatment (A group + B group) but only 50 have this parameter determined both at the beginning and end of the period.
  61 patients ended the period of 7 weeks of placebo treatment (A group + B group) but only 50 have this parameter determined both at the beggining and at the end of the period.
Measure: Mean (95% Confidence Interval); unit: % (FEV1)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 50 | 50
% (FEV1) | 4.1 [0.0 to 8.3] | 4.3 [0.1 to 8.5]

2. Secondary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Forced Vital Capacity (FVC)
Description: Changes from baseline on measurements of respiratory function defined by forced vital capacity (FVC).
  Mean difference between 7 weeks after treatment visit and baseline visit is registered.
Time Frame: 7 weeks
Population: 59 patients ended the period of 7 weeks of liraglutide treatment (A group + B group) but only 50 have this parameter determined both at the beginning and end of the period.
  61 patients ended the period of 7 weeks of placebo treatment (A group + B group) but only 50 have this parameter determined both at the beginning and end of the period.
Measure: Mean (95% Confidence Interval); unit: % (FVC)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 50 | 50
% (FVC) | 5.4 [2.1 to 8.7] | 0.2 [-2.5 to 3.1]

3. Secondary Outcome: Changes From Baseline in Serum Levels of Surfactant A and D Protein
Description: Changes from baseline in serum levels of surfactant A and D protein. Values for surfactant A or D protein after 7 treatment weeks (liraglutide or placebo) are registered.
Time Frame: 7 weeks
Population: 59 patients ended the period of 7 weeks of liraglutide treatment (A group + B group) but only 48 have this parameter determined both at the beginning and end of the period.
  61 patients ended the period of 7 weeks of placebo treatment (A group + B group) but only 48 have this parameter determined both at the beginning and end of the period.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 48 | 48
ng/ml
  A protein | 40.9 [30.8 to 44.5] | 41.3 [21.5 to 50.3]
  D protein | 169.6 [108.1 to 233.6] | 201.5 [115.3 to 284.7]

4. Secondary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Maximum Mid-expiratory Flow (FEF25-75)
Description: Changes from baseline on measurements of respiratory function defined by Maximum mid-expiratory flow (FEF25-75).
  Mean difference between 7 weeks after treatment visit and baseline visit is registered.
Time Frame: 7 weeks
Population: 59 patients ended the period of 7 weeks of liraglutide treatment (A group + B group) but only 46 have this parameter determined both at the beginning and end of the period.
  61 patients ended the period of 7 weeks of placebo treatment (A group + B group) but only 46 have this parameter determined both at the beginning and end of the period.
Measure: Mean (95% Confidence Interval); unit: % (FEF25-75)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 46 | 46
% (FEF25-75) | 8.0 [-4.1 to 20.1] | 12.5 [2.2 to 22.8]

5. Secondary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Forced Expiratory Volume in 1 Second/Forced Vital Capacity (FEV1/FVC)
Description: Changes from baseline on measurements of respiratory function defined by forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC).
  Mean difference between 7 weeks after treatment visit and baseline visit is registered.
Time Frame: 7 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: % (FEV1/FVC)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 50 | 50
% (FEV1/FVC) | -2.1 [-5.1 to 0.9] | 1.7 [-0.8 to 4.2]

6. Secondary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Residual Volume (RV)
Description: Changes from baseline on measurements of respiratory function defined by residual volume (RV).
Time Frame: 7 weeks
Population: 59 patients ended the period of 7 weeks of liraglutide treatment (A group + B group) but only 12 have this parameter determined both at the beginning and end of the period.
  61 patients ended the period of 7 weeks of placebo treatment (A group + B group) but only 12 have this parameter determined both at the beginning and end of the period.
Measure: Mean (95% Confidence Interval); unit: % (RV)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 12 | 12
% (RV) | 3.2 [-17.5 to 24.1] | -1.1 [-25.4 to 23.1]

7. Secondary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Total Lung Capacity (TLC)
Description: Changes from baseline on measurements of respiratory function defined by Total lung capacity (TLC).
Time Frame: 7 weeks
Measure: Mean (95% Confidence Interval); unit: % (TLCO)
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 12 | 12
% (TLCO) | -2.6 [-11.9 to 6.6] | -3.1 [-9.5 to 3.2]

8. Secondary Outcome: Changes From Baseline on Measurements of Respiratory Function Defined by Residual Functional Capacity (RFC)
Description: Changes from baseline on measurements of respiratory function defined by Residual functional capacity (RFC) are registered.
  However, this parameter was not determined in patients due to an error in the programm used.
Time Frame: 7 weeks
Population: This parameter was not determined in patients due to an error in the programm used.
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 weeks of treatment.
Arm/Group | Liraglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/70
Other Adverse Events (participants affected / at risk) | 19/70 | 13/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=70) | Placebo (N=70)
Ischemic stroke (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=70) | Placebo (N=70)
Gastrointestinal disorders (Gastrointestinal disorders) | 19 (20) | 4 (4)
Infections and infestations (Infections and infestations) | 1 (1) | 3 (3)
Nervous system disorders (Nervous system disorders) | 2 (2) | 2 (2)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2) | 1 (1)
General disorders and administration site conditions (General disorders) | 2 (2) | 0 (0)
Cardiac disorders (Cardiac disorders) | 1 (1) | 1 (1)
Traumatic injuries, poisonings and complications of therapeutic procedures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Congenital, family and genetic disorders (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02889510/Prot_SAP_000.pdf